CLINICAL TRIAL: NCT00508677
Title: Mazindol in Children With Attention Deficit Hyperactivity Disorder Design Study to Explore the Effectiveness, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Two Orally Administered Doses of Mazindol.
Brief Title: Mazindol in Children With ADHD : Open-label, Efficacy, Safety and Pharmacokinetic Pilot Trial
Acronym: MAZDAH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick VACHER, Department Clinical Research of Developpement
Other Study IDs: P060104
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2007-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Mazindol
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective pilot trial will evaluate the efficacy, safety, tolerability and pharmacokinetic (PK) and pharmacodynamic (PD) properties of mazindol.

DETAILED DESCRIPTION:
The most common intervention for Attention Deficit Hyperactivity Disorder (ADHD) is pharmacological treatment with methylphenidate (MPH). Effects of MPH on ADHD symptoms in children is extremely well-informed. Mazindol is a psychostimulant and a wake-promoter agent which may have similar actions to MPH in the central nervous system. However, there is no record of the effects, safety, tolerability of Mazindol in children with ADHD. Mazindol (dose 0.5 or 1.0 mg/day) should prove to be useful in the treatment of ADHD symptoms in children. Based on clinical assessments and serum concentrations after oral administration of mazindol to children (6-12 years) with ADHD, this prospective pilot trial will evaluate the efficacy, safety, tolerability and pharmacokinetic (PK) and pharmacodynamic (PD) properties of mazindol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects can be boys or girls
* Subjects must be aged between 6 to 12 years,
* Tanner 1 ou 2
* Subjects with a diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Diseases, Fourth Edition (DSM-IV) criteria
* ADHD-RS score of ≥ 31 as determined by investigator at screening visit.
* Drug free including psychostimulants (10 days before the screening visit)
* Informed Consent Form signed by the subject and both parents
* Healthy on the basis of a physical examination, medical history and the results of blood hematology tests.

Exclusion Criteria:

* Any clinically unstable psychiatric condition including, but not limited to the following: acute mood disorder, bipolar disorder, obsessive-compulsive disorder (OCD), autism or Asperger…
* Sleep Disorders including narcolepsy, hypersomnia (according to International Classification of Sleep Disorders (ICSD) criteria
* Chronic diseases (e.g. asthma…)
* Current eating disorder (e.g. bulimia, anorexia nervosa) or history of an eating disorder during infancy
* Mental retardation (IQ < 80)
* Hyperthyroidism
* Subjects with history of seizures, glaucoma or familial hypertension
* Heart pathologies

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: childrens
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric KONOFAL, MD-PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Robert Debre, Paris, France